CLINICAL TRIAL: NCT01443052
Title: Study of the Temporospatial Gait Parameters With the Electronic Carpet "GAITRite" in Patients With Walking Impairment After Stroke and in Old Faller Subjects
Brief Title: Gait Parameters Analysis in Post-stroke Patients and in Elderly Fallers
Acronym: GAITRITE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: UC1002
Record Dates: First submitted 2011-05-04; First posted 2011-09-29 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Healthy; Thalamic Pain Syndrome; Fallers
Keywords: Gait stability; Spatiotemporal parameters; Walking; Elderly people; Stroke; Fallers
MeSH Terms: conditions — Thalamic Diseases; Stroke | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- post-stroke patients: Stroke patients who had only one cerebrovascular accident, at least one year before inclusion and Able to walk without using assisting devices or ambulatory aids
  Interventions: Other: Gait analysis
- healthy subjects: Aged 65 to 80 years
  Interventions: Other: Gait analysis
- fallers: Reported 2 or more falls within 6 months prior to the beginning of the study and Able to walk without using assisting devices or ambulatory aids
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — walking on an electronic walkway GAITRite® at self-selected speed

SUMMARY:
A large proportion of falls in older people occurs when walking. Most studies have recently demonstrated correlation between the variations in spatiotemporal gait parameters and fall risk in elderly and in several diseases. The investigators objective is to analyse this parameters in population with gait stability disorders (post-stroke patients and fallers) to identify the most valuable and to develop/test a conglomerate stability score.

DETAILED DESCRIPTION:
Temporal-spatial gait parameters will be recorded in subjects aged 65-80 years : 30 healthy people, 30 patients at least one year post-stroke, and 30 fallers while walking on an electronic walkway GAITRite® at self-selected speed.

ELIGIBILITY:
1. For healthy subjects

   * Aged 65 to 80 years (included) ;
   * Patient has been informed and has signed the consent form.
2. For post-stroke patients

   * Aged 65 to 80 years (included) ;
   * Stroke patients who had only one cerebrovascular accident, at least one year before inclusion ;
   * Able to walk without using assisting devices or ambulatory aids ;
   * No cardiovascular contraindication ;
   * No history of neurological diseases with influence on walking capacities (excepted stroke) ;
   * No history of vestibular or orthopaedic (lower limb) disorders ;
   * No amblyopia ;
   * Patient has been informed and has signed the consent form.
3. For fallers

   * Aged 65 to 80 years (included) ;
   * Reported 2 or more falls within 6 months prior to the beginning of the study ;
   * Able to walk without using assisting devices or ambulatory aids ;
   * No cardiovascular contraindication ;
   * No history of neurological diseases with influence on walking capacities ;
   * No history of vestibular or orthopaedic (lower limb) disorders ;
   * No amblyopia ;
   * Patient has been informed and has signed the consent form.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: subjects aged 65-80 years : 30 healthy people, 30 patients at least one year post-stroke, and 30 fallers
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
GAIT parameters | at inclusion
  Spatiotemporal gait parameters registered by a GAITRite walkway system, including mean and coefficient of variation for step and cycle length and time, base of support, speed, cadence, single and double support phase, stance and swing phase.

SECONDARY OUTCOMES:
Functional Ambulation Performance Score | at inclusion
  a score which represents a quantification of patients' gait based on a selection of spatiotemporal parameters obtained at a self-selected speed.
Rivermead Motricity Index | at inclusion
  For post-stroke patients
Berg Balance Scale | at inclusion
  For post-stroke patients

CONTACTS AND LOCATIONS:
Overall Officials: Alain Yelnik, Principal Investigator — PRM department
Locations (1):
- PRM Department - Lariboisiere Hospital, Paris, France

REFERENCES:
- [Background] Hausdorff JM, Rios DA, Edelberg HK. Gait variability and fall risk in community-living older adults: a 1-year prospective study. Arch Phys Med Rehabil. 2001 Aug;82(8):1050-6. doi: 10.1053/apmr.2001.24893. PMID 11494184
- [Background] Hausdorff JM, Nelson ME, Kaliton D, Layne JE, Bernstein MJ, Nuernberger A, Singh MA. Etiology and modification of gait instability in older adults: a randomized controlled trial of exercise. J Appl Physiol (1985). 2001 Jun;90(6):2117-29. doi: 10.1152/jappl.2001.90.6.2117. PMID 11356774
- [Background] Bilney B, Morris M, Webster K. Concurrent related validity of the GAITRite walkway system for quantification of the spatial and temporal parameters of gait. Gait Posture. 2003 Feb;17(1):68-74. doi: 10.1016/s0966-6362(02)00053-x. PMID 12535728
- [Background] Menz HB, Latt MD, Tiedemann A, Mun San Kwan M, Lord SR. Reliability of the GAITRite walkway system for the quantification of temporo-spatial parameters of gait in young and older people. Gait Posture. 2004 Aug;20(1):20-5. doi: 10.1016/S0966-6362(03)00068-7. PMID 15196515
- [Background] Balasubramanian CK, Neptune RR, Kautz SA. Variability in spatiotemporal step characteristics and its relationship to walking performance post-stroke. Gait Posture. 2009 Apr;29(3):408-14. doi: 10.1016/j.gaitpost.2008.10.061. Epub 2008 Dec 3. PMID 19056272
- [Background] Gouelle A, Megrot F, Presedo A, Pennecot GF, Yelnik A. Validity of Functional Ambulation Performance Score for the evaluation of spatiotemporal parameters of children's gait. J Mot Behav. 2011;43(2):95-100. doi: 10.1080/00222895.2010.538768. PMID 21298587